CLINICAL TRIAL: NCT06067334
Title: Complete Digital Workflow for Construction of Full Arch Implant Supported Screw Retained Restoration: Accuracy of Different Impressions Techniques on Implant and Abutment Levels (Cross-over Study)
Brief Title: Complete Digital Workflow for Construction of Full Arch Implant Supported Screw Retained Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Fatma mahanna, lecturer of prosthodontics, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: J0104023RP
Record Dates: First submitted 2023-09-25; First posted 2023-10-04 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Accuracy
Keywords: Accuracy; implant level impression; abutment level impression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Open tray impression technique) (Active Comparator): After osseointegration, a conventional open tray splinted impression technique will be made for each patient on the implant/abutment level.
  Interventions: Other: full arch implant supported screw retained restoration with conventional impression technique
- Digital impression (Active Comparator): Scan bodies implant level/abutment level will be tightened for each patient, and a digital intraoral scanner will be used to scan the scan bodies for making implant level/abutment level digital impressions.
  Interventions: Other: full arch implant supported screw retained restoration with conventional digital technique

INTERVENTIONS:
Other: full arch implant supported screw retained restoration with conventional impression technique — surgical procedures: Implant installation Prosthetic procedures: Conventional impression fabrication of full arch implant supported screw-retained restoration evaluation: Accuracy, Passive fit
  Arms: Conventional (Open tray impression technique)
Other: full arch implant supported screw retained restoration with conventional digital technique — surgical procedures: Implant installation Prosthetic procedures: Digital impression fabrication of full arch implant-supported screw-retained restoration evaluation: Accuracy, Passive fit
  Arms: Digital impression

SUMMARY:
aim: to compare the accuracy of the conventional and digital impression when will be performed on implant level or abutment level in Complete digital workflow for construction of full arch implant supported screw-retained restoration.

DETAILED DESCRIPTION:
The patient will be selected according to the following criteria:

1. Free from any systemic disease that may interfere with proper Osseointegration of implants, which will be assessed by thorough medical investigations.
2. Patients having completely edentulous maxilla and mandible for at least 6 months after the last extraction.
3. Normal maxilla mandibular relationship with adequate inter-arch space, measured by tentative jaw relation.
4. Sufficient residual alveolar ridge.

Exclusion criteria include:

1. Local or general contraindications for surgical procedures.
2. Patients with TMJ disorders or poor neuromuscular coordination or parafunctional habits.
3. Severe inter-maxillary skeletal discrepancy or limited inter-arch space.
4. Heavy smokers.

   * For all patients, conventional complete dentures are constructed.
   * Implants installed in the edentulous maxilla and mandible in each target position guided by stereolithographic stent. A delayed loading protocol is followed in this study.
   * After osseointegration, a conventional open tray splinted impression technique will be made for each patient on the implant/abutment level.
   * Scan bodies' implant level/abutment level will be tightened for each patient, and a digital intraoral scanner will be used to scan the scan bodies for making implant level/abutment level digital impressions.

Accuracy will be evaluated as follows:

* 3D inspection software using the best-fit alignment algorithm will be utilized to calculate the 3D deviation of each impression using the root mean square (RMS) error.
* Passive fit of the framework will be evaluated at the time of insertion.

ELIGIBILITY:
Inclusion Criteria:

* Free from any systemic disease that may interfere with proper Osseointegration of implants, which will be assessed by thorough medical investigations.
* Patients having completely edentulous maxilla and mandible for at least 6 months after the last extraction.
* Normal maxilla mandibular relationship with adequate inter-arch space as verified by tentative jaw relation.
* Sufficient residual alveolar ridge.

Exclusion Criteria:

* Local or general contraindications for surgical procedures.
* Patients with TMJ disorders or poor neuromuscular coordination or parafunctional habits.
* Severe inter-maxillary skeletal discrepancy or limited inter-arch space.
* Heavy smokers.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Best fit alignment to calculate 3D deviation of each impression | 3 months
  3D inspection software (Geomagic Control X) using the best-fit alignment algorithm will be utilized to calculate the 3D deviation of each impression using the root mean square (RMS) error.

SECONDARY OUTCOMES:
Passive fit | 3 months
  Passive fit of framework will be evaluated at time of insertion (Sheffield test)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gamal, MD, Principal Investigator — Mansoura university, faculty of dentistry
Locations (1):
- Faculty of dentistry, mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No